CLINICAL TRIAL: NCT05039268
Title: A Phase 2 Open Label Trial of 3K3A-APC in Amyotrophic Lateral Sclerosis
Brief Title: 3K3A-APC for Treatment of Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Macquarie University, Australia (Other)
Collaborators: ZZ Biotech, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZZ-3K3A-202
Record Dates: First submitted 2021-08-23; First posted 2021-09-09 (Actual); Results first posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2022-09

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Amyotrophic Lateral Sclerosis; MND; Motor Neurone Disease; 3K3A-APC
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — 3K3A-APC protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 15mg Dose Group (Active Comparator): Participants will receive a fixed dose regimen of five doses of 15mg.
  Interventions: Drug: 3K3A-APC Protein
- 30mg Dose Group (Active Comparator): Participants will receive a fixed dose regimen of five doses of 30mg.
  Interventions: Drug: 3K3A-APC Protein

INTERVENTIONS:
Drug: 3K3A-APC Protein — 3K3A-APC with intravenous dosing of five doses of either 15mg or 30mg at 12 hourly interval. The first 8 patients will receive 15mg dose, and the next 8 patients will receive 30mg dose.
  Other Names: 3K3A-APC

SUMMARY:
Phase 2 open label trial to investigate the safety and potentially efficacy of 3K3A-APC in patients with Amyotrophic Lateral Sclerosis (ALS).

DETAILED DESCRIPTION:
This Phase 2 open label trial seeks to investigate whether a novel therapy named 3K3A-APC is safe and potentially effective in patients with Amyotrophic Lateral Sclerosis (ALS). A total of 16 patients with ALS will be enrolled into 2 dose cohorts with five doses of 15mg or 30mg doses given 12 hours apart in each cohort. The primary study outcomes are to ensure the safety and tolerability of 3K3AAPC in ALS patients, and to determine whether 3K3A-APC is able to reduce the pathological changes that might possibly cause ALS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have clinically definite ALS (Awaji Criteria)
2. Male or female age 18 years and less than 75 years at time of ALS study
3. Symptom onset less than 36 months before screening
4. Diagnosis of ALS less than 24 months before screening
5. Clinically definite Upper Motor Neuron signs

Exclusion Criteria:

1. Current treatment with anticoagulants (e.g., warfarin, novel oral anticoagulants, heparin) that might preclude safe completion of the lumbar puncture
2. Condition that precludes the safe performance of routine lumbar puncture, such as prohibitive lumbar spinal disease, bleeding diathesis, or clinically significant coagulopathy or thrombocytopenia
3. Use of investigational drugs or devices within 60 days prior to Baseline (dietary supplements taken outside of a clinical trial are not exclusionary, e.g., coenzyme Q10)
4. Prolonged prothrombin time or activated partial thromboplastin time >2xULN
5. Severe hypertension or hypotension
6. Glomerular filtration rate (GFR) <35 mL/min
7. Forced vital capacity (FVC) at screening of <50% of predicted
8. Prior exposure to any exogenous form of APC
9. Inability to lie flat for procedures (MRI, PET, LP)
10. Pregnant or lactating during the study period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Rowe, PhD, MD, Principal Investigator — Macquarie University, Australia
Locations (1):
- Macquarie University, Macquarie Park, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 15mg Dose Group | 30mg Dose Group
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 15mg Dose Group | 30mg Dose Group | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Full Range); unit: years] | 59.5 [42 to 73] | 57.1 [39 to 71] | 58.3 [39 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 8 | 8 | 16
ALSFRS-R Score [Mean (Full Range); unit: units on a scale] — ALSFRS-R measures 12 aspects of physical function, ranging from subject's ability to swallow and use utensils to climbing stairs and breathing. Each function is scored from 4 (normal) to 0 (no ability). The maximum score is 48 and the minimum is 0.
  units on a scale | 30.875 [19 to 45] | 37.125 [20 to 46] | 34.0 [19 to 46]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Any Serious Adverse Events or Any Adverse Events With Severity Higher Than "Moderate".
Description: Number of participants who had any serious adverse events or any adverse events with severity higher than "moderate", as determined by the Principal Investigator, using the composite safety assessment including clinical laboratory testing (full blood count, biochemistry, coagulation, iron study, CSF analysis and ECG), physical examination and self-reporting of adverse events. All clinical significant findings in the composite safety assessment were reported as adverse events.
Time Frame: 15 Days
Population: All dosed participants are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 15mg Dose Group | 30mg Dose Group
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

2. Primary Outcome: Percentage of Change in PERSI Score in the Motor Cortex Before and After Dosing
Description: PERSI (Parametric Estimation of Reference Signal Intensity) score is the measurement of microglial activation in the motor cortex utilising serial [18F]FEMPA PET imaging. The percentage of change in PERSI score before and after dosing in the two (2) dose cohorts is calculated.
Time Frame: 7 Days
Population: In total, 8 participants were included in the data analysis, with 5 participants in the 15mg group and 3 participants in the 30mg group.
Measure: Mean (Full Range); unit: Percentage of change
Arm/Group | 15mg Dose Group | 30mg Dose Group
Number analyzed (Participants) | 5 | 3
Percentage of change | -0.14 [-4.01 to 2.63] | 0.53 [-0.96 to 2.61]

3. Secondary Outcome: Diffusion Kurtosis Using MRI Scan
Description: Change in diffusion kurtosis using MRI scan of the brain to determine whether the blood brain barrier integrity can be measured in ALS by Magnetic Resonance Imaging, and whether 3K3A-APC is able to repair it
Time Frame: 7 Days
Reporting Status: Not Posted

4. Secondary Outcome: Monocyte Activation
Description: Change in the level of monocyte activation in the peripheral blood utilising a novel method.
Time Frame: 7 Days
Reporting Status: Not Posted

5. Secondary Outcome: Cytokine Level
Description: Change in cytokine level in serum, plasma and CSF.
Time Frame: 7 Days
Reporting Status: Not Posted

6. Secondary Outcome: Chemokine Level
Description: Change in chemokine level in serum, plasma and CSF.
Time Frame: 7 Days
Reporting Status: Not Posted

7. Secondary Outcome: Neurofilament Level
Description: Change in neurofilament level in serum, plasma and CSF.
Time Frame: 7 Days
Reporting Status: Not Posted

8. Secondary Outcome: Soluble CD14 Level
Description: Change in soluble CD14 level in serum, plasma and CSF.
Time Frame: 7 Days
Reporting Status: Not Posted

9. Secondary Outcome: Kynurenine Level
Description: Change in kynurenine level in serum, plasma and CSF.
Time Frame: 7 Days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Day-of-consent through end-of-participation, 15 days
Description: Adverse events are continuously collected from day-of-consent through end-of-participation for each participant.
Arm/Group | 15mg Dose Group | 30mg Dose Group
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 6/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 15mg Dose Group (N=8) | 30mg Dose Group (N=8)
Fall (Injury, poisoning and procedural complications) | 2 | 1
Headache (Nervous system disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 0 | 2
Neutrophilia (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Blood calcium increased (Investigations) | 1 | 0
Blood bicarbonate increased (Investigations) | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Catheter site extravasation (General disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The main limitation of the study is the small number of participants in the [18F]FEMPA PET analysis, which is one of the primary outcomes. In total, only 8 participants (5 in the 15mg group and 3 in the 30mg group) were analysed. The reasons for not including in the analysis are: PET scan data loss due to technical issues (1 participant), PET scan not being performed due to FEMPA production/QC failure (1 participant), and data being uninterpretable at analysis stage (6 participants).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/68/NCT05039268/Prot_SAP_000.pdf